CLINICAL TRIAL: NCT03643822
Title: Adjuncts for Adductor Block: Dexamethasone,Dexmedetomidine, or Combination to Reduce Pain. A Randomized Controlled Comparison of the Analgesic Effects Following ACL Repair
Brief Title: Adjuncts for Adductor Block: Dexamethasone,Dexmedetomidine, or Combination to Reduce Pain
Acronym: AADDCToR
Status: Recruiting | Phase: Phase 4 | Type: Interventional
Sponsor: Women's College Hospital (Other)
Collaborators: University Health Network, Toronto (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Factorial | Masking: Double | Purpose: Other
Other Study IDs: 2018-0164-B
Record Dates: First submitted 2018-06-25; First posted 2018-08-23 (Actual); Last update posted 2025-03-27 (Actual); Status verified 2025-03

CONDITIONS: ACL Injury
Keywords: ACB adjuncts; Dexamethasone; Dexmedetomidine; post operative analgesia
MeSH Terms: conditions — Anterior Cruciate Ligament Injuries | interventions — Dexamethasone; Dexmedetomidine; Sodium Chloride

STUDY DESIGN:
Intervention Model Description: There will be prospective,randomized,controlled,parallel group,factorial,1:1:1:1 allocation,operator,patient and assessor blinded clinical trial.
Who Masked: Participant, Outcomes Assessor
Masking Description: Patients who give written informed consent will be randomly assigned on the day of surgery to either of the four study groups using a computer-generated block randomization schedule in blocks of varying sizes. Group allocation will not be disclosed to the anesthesiologist performing the ACB. An anesthesia assistant will receive an opaque envelope containing the result of randomization, and will prepare the block study solution in identical syringes. The patient receiving ACB will also be blinded to the study solution injected. Furthermore, outcome assessment will be performed by a blinded research assistant.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (4):
- Dexamethasone vs. Control comparison (Active Comparator): Freezing + dexamethasone(4mg)+1 ml of saline
  Interventions: Drug: Dexamethasone 4mg; Other: Saline
- Dexmedetomidine vs. Control comparison (Active Comparator): Freezing + dexmedetomidine(50ug) + 1.5 ml of saline
  Interventions: Drug: Dexmedetomidine; Other: Saline
- Dexamethasone and Dexmedetomidine (Active Comparator): Freezing+dexamethasone(4mg)+dexmedetomidine(50ug) + 0.5 ml of saline
  Interventions: Drug: Dexamethasone 4mg; Drug: Dexmedetomidine; Other: Saline
- Control Group-Placebo (Sham Comparator): Freezing + 2ml saline
  Interventions: Other: Saline

INTERVENTIONS:
Drug: Dexamethasone 4mg — To guarantee rapid onset as well as effective postoperative analgesia, a 20 mL volume of local anesthetic has been selected for performing the ACB. The block solution will be a 20 ml volume for all groups, prepared by mixing 18 ml of ropivacaine 0.5% mixed with an additional 2 ml prepared according to the randomization.
  Other Names: Preservative free Dexamethasone
  Arms: Dexamethasone and Dexmedetomidine; Dexamethasone vs. Control comparison
Drug: Dexmedetomidine — To guarantee rapid onset as well as effective postoperative analgesia, a 20 mL volume of local anesthetic has been selected for performing the ACB. The block solution will be a 20 ml volume for all groups, prepared by mixing 18 ml of ropivacaine 0.5% mixed with an additional 2 ml prepared according to the randomization.
  Other Names: Dexmedetomidine Hydrochloride 0.5 MG/ML
  Arms: Dexamethasone and Dexmedetomidine; Dexmedetomidine vs. Control comparison
Other: Saline — Control/Placebo intervention

SUMMARY:
The aim of this multi-centered study is to evaluate the effects of two distinct Adductor Canal Block (ACB) adjuncts, dexamethasone and dexmedetomidine, and their combination, on postoperative analgesia in patients undergoing Anterior Cruciate Ligament (ACL) Repair.

DETAILED DESCRIPTION:
Anterior cruciate ligament repair (ACLR) is a surgical procedure of the knee associated with moderate to severe postoperative pain lasting beyond 24 hours following surgery. Provision of adequate postoperative analgesia is a prerequisite for performing this procedure on outpatient basis. By virtue of their analgesic effects, peripheral nerve blocks (PNBs), such as adductor canal block (ACB), have thus become part of the care standard for this surgical procedure.

Though ACB provides effective pain relief, the duration of analgesia associated with this block is limited to eight hours postoperatively. As a result, patients having outpatient ACLR may experience severe pain following discharge, require additional opioid analgesics to control their pain, and even visit the emergency department for acute pain management. Consequently, perioperative care for the young outpatient population undergoing this procedure is an area where improvement is needed.

Mixing adjuncts with local anesthetics can prolong the duration of analgesia of PNBs; both dexmedetomidine and dexamethasone have been shown to effectively extend the duration of PNB analgesia by 60% and 80% hours, respectively. The use of dexamethasone is wide spread, and dexmedetomidine is progressively gaining popularity.

At Toronto Western Hospital, the use of adjuncts is left to the discretion of the anesthesiologists administering PNB; and dexamethasone is occasionally used to prolong block duration. The alternative approach to prolonging block duration is using ambulatory ACB catheters, but this is an expensive option that is applicable to select patients, and it is not available at the TWH.

Importantly, these adjuncts seem to exert their effect through independent mechanisms; thus there may be an advantage to combining adjuncts together. Further prolongation of the duration of analgesia is desirable, as the prolongation of block duration associated with each of these two adjuncts, alone, falls short of the duration of worst postoperative pain following ACLR. Consequently, the investigators aimed to explore whether the combination of these two adjuncts offers an incremental benefit over either of them alone, by examining their potential additive or synergistic effect.

This randomized controlled trial compares the effect of using perineural dexamethasone, dexmedetomidine, and their combination to Control on the duration of postoperative analgesia in patients having ambulatory ACLR with ACB.

ELIGIBILITY:
Inclusion Criteria:

* English Speaking
* ASA 1-3 patients
* BMI <40

Exclusion Criteria:

* Refusal or inability to provide informed consent
* Any contraindication to regional anesthesia including coagulopathy or bleeding diathesis, allergy to local anesthetics, infection, nerve injury or malignancy at the site of the block
* History of alcohol/drug dependence
* History of long term opioid intake or chronic pain disorder
* History of preexisting neuropathy in the operative leg
* History of significant psychiatric conditions that may affect patient assessment
* Inability to understand the informed consent and demands of the study
* Allergy to any of the components of the multimodal analgesic regimen
* Revision of ACL repair
* Diabetes
* Significant bradycardia (baseline heart rate ≤ 40 beats per minute)

Ages: 18 Years to 50 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 252 (Estimated)
Dates: Start 2020-02-21 (Actual); Primary Completion 2026-12 (Estimated); Study Completion 2026-12 (Estimated)

PRIMARY OUTCOMES:
Oral opioid consumption | time of the block to 24 hours after
  Cumulative 24 hour oral morphine equivalent consumption

SECONDARY OUTCOMES:
Intra-operative opioid consumption | Duration of surgery: From start of surgery (defined as anesthesia start) to end of surgery (defined as anesthesia end)
  Cumulative intra-operative opioid consumption in morphine equivalent
PACU opioid consumption | From time of arrival (hh:mm) in PACU to time of PACU discharge (hh:mm) assessed up to 24 hours
  Cumulative oral morphine equivalent consumption during time stayed in PACU
Time to first analgesic request in PACU | From time of arrival in PACU (hh:mm) up to time of PACU discharge (hh:mm) assessed in minutes up to 24 hours ((e.g. patient arrives in PACU 12:00 then patient is given first pain medication in PACU at 12:30; Time to first analgesic request = 30 min)
  The time (hh:mm) first pain medication given in PACU
Time to PACU discharge | From time of arrival (hh:mm) in PACU to time discharged (hh:mm) from PACU assessed in minutes (e.g. patient arrives in PACU 12:00 then patient discharged from PACU 12:30; Time to PACU discharge = 30 min)
  how fast patient recovered and discharged from PACU (measured in minutes)
Visual Analogue Scale-Pain scores - minimum score = 0 and maximum score = 10 | discharge from hospital to 2 days after surgery
  pain scores at 0, 2, 4, 6, 12, 24, 36, and 48 hours postoperatively
Opioid consumption | discharge from hospital to 2 days after surgery
  analgesic consumption at 6, 12, 24, 36, and 48 hours postoperatively
Risk of block-related complications | one week post operatively
  adverse symptoms related to the block
Risk of opioid-related side effects | two week post operatively
  adverse symptoms related to oral pain medication consumption
Quality of recovery-15 (QoR15) (0-10, where 0 = none of the time [poor] and 10 = all of the time [excellent] | discharge from hospital to 24 hours after surgery
  measured using the Quality of recovery-15 at 12 and 24 hours postoperatively
Time to hospital discharge | From time of end of surgery [(hh:mm) defined as anesthesia end] up to time of hospital discharge (hh:mm) assessed in minutes up to 24 hours (e.g. surgery ends 12:00, then patient discharged from the hospital at 13:00; Time to hospital discharge = 60min
  Measures of recovery (how many minutes from end of surgery to discharge from hospital)
Time to first analgesic request at home (after discharge) | discharge from hospital to 24 hours after surgery
  first time(hh:mm) patient took an oral pain medication
Visual Analogue Scale-Satisfaction scores - where 0 = not satisfied and 10 = very satisfied | evaluated at 12 and 24 hours post-surgery
  A visual analogue scale used to measure how satisfied the study participant is with the pain relief received for shoulder surgery
Presence/absence of nerve block complications | time from block onset to 2 days,2 weeks after surgery
  adverse symptoms related to the block

CONTACTS AND LOCATIONS:
Overall Officials: Richard Brull, MD, Principal Investigator — Women's College Hospital
Locations (1):
- Women's College Hospital, Toronto, Ontario, Canada